CLINICAL TRIAL: NCT01768039
Title: Randomised Double Blind Placebo-controlled Trial of Vitamine D Supplement in Multiple Sclerosis
Brief Title: Vitamine D in Multiple Sclerosis
Acronym: MSVit
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mahmoud Abedini, associate professor of neurology, Mazandaran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS-1191
Record Dates: First submitted 2013-01-11; First posted 2013-01-15 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Vitamin D; EDSS; ARR
MeSH Terms: conditions — Multiple Sclerosis | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Active Comparator): treatment with weekly 50000IU vitamin D
  Interventions: Drug: Vitamin D
- Placebo (Placebo Comparator): Treatment with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D
  Arms: Vitamin D
Drug: Placebo
  Arms: Placebo

SUMMARY:
Two hundred and forty patients with multiple sclerosis who met the study criteria will be enrolled in this randomized double blind placebo-controlled clinical trial.

They will randomly assigned to placebo or vitamin D treatment group. The total time of study is 52 weeks and the vitamin D group will be treated by weekly 50000 International unit(IU) vitamin D, while the other group will receive weekly placebo. The annual relapse rate and EDSS will be compared at baseline, month 6 and 12.

ELIGIBILITY:
Inclusion Criteria:

* BMI:18-30kg/m2
* caucasian race
* Relapsing remitting multiple sclerosis
* treatment with interferon beta

Exclusion Criteria:

* Recent vitamin D supplement therapy
* Restricted fat diet
* nephrolithiasis in recent 5 years
* Past history of hyperparathyroidism, sarcoidosis, cancer
* Past history of hepatic disease
* Past history of gastrointestinal disease
* Past history of mycobacterial infection
* Past history of hypercalcemia and hypercalciuria
* serum creatinine>1.5
* Smoking, drug abuse and corticosteroid therapy in recent year
* treatment with thiazides or other drugs that inhibit vitamin D absorption
* Disease attack in recent 2 months
* Serum Ca>2.6mm0l/L
* Serum 25(OH)D>85mmol/L
* hypersensitivity to cholecalciferol
* Past history of heart disease
* Major depression
* Uncontrolled hypertension (BP>180/110)
* Immunosuppressive therapy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-08 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Expanded disability state scale score (EDSS) | Changes in EDSS from baseline to 6 months

SECONDARY OUTCOMES:
Annual relapse rate(ARR) | Changes in ARR from baseline to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mazandaran University of medical sciences, Sari, Mazandaran, Iran